CLINICAL TRIAL: NCT05619679
Title: A Clinical Practice Snapshot on Pediatric Kidney Transplantation Healthcare in Europe
Brief Title: A Clinical Practice Snapshot on Pediatric Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PKT.Clinical.Snapshot
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplant Failure
Keywords: Kidney transplantation
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Kidney Transplantation — Kidney transplantation

SUMMARY:
The aim is to create an overview of the similarities and differences in daily practice among the different centers performing pediatric kidney transplantation in Europe.

For this purpose, a Clinical Practice Snapshot will be used to provide insight in the current approaches.

DETAILED DESCRIPTION:
In order to create an overview of the current care for pediatric kidney transplant (PKT) recipients a clinical practice snapshot was developed.

All participating centers were asked to answer 6 clinical questions on their last 30 transplanted patients.

Patient characteristics, donor charactertistics, use of stents, immunosuppressive medication and renal function are compared between centers.

ELIGIBILITY:
Inclusion Criteria:

* Kidney received <18 years
* at least one month of follow-up
* transplantation and follow-up in dedicated PKT center

Exclusion Criteria:

* combined transplantation

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All pediatric kidney recipients that were transplanted in one of the participating centers and followed up for at least one month
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Graft survival | at end of follow-up at least one month
  Functioning graft
Donor type | At transplantation
  Living or deceased donor

SECONDARY OUTCOMES:
Immunosuppressants prescribed at discharge | 2 weeks
  Immunosuppressive medication at discharge after transplant
Number of infections | end of follow-up, at least one month
  Viral infections after transplantations

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Researchers from centers that contributed can request anonymized data
Supporting Information: ICF